CLINICAL TRIAL: NCT02710448
Title: May Metformin be Used in Renal Failure?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI11-PR-LALAU-2; 2012-001207-20 (EudraCT Number)
Record Dates: First submitted 2012-08-10; First posted 2016-03-16 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Renal Disorder Associated With Type II Diabetes Mellitus
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): Metformin in patients with renal failure
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin (Glucophage ®), oral antidiabetic, will be administered as it is usually recommended: engaged during or at the end of the meal in the evening for the single dose 500 mg (Phase 1), the evening and morning for total doses of 1000 mg, 2000 mg and 3000 mg (with, respectively, 2 tab. 500 mg, 2 tab. to 1000 mg, 1 tab. to 1000 mg and 2 tab. to 1000 mg), a fourth dose is also scheduled to stage one (3000 mg / d)
  Other Names: phase1 : 500 mg/d; phase2 : 2 x 500 mg/d; phase3 : 2 x 1000 mg/d; phase4 : 3 x 1000 mg/d

SUMMARY:
The study is to treat metformin dose-escalation diabetic subjects of all stages of renal failure (stages 1-5) and compare their rates of erythrocyte metformin (best reflections of a possible accumulation than those of plasma) to the therapeutic range. A number of 12 patients by stage is considered, 60 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients not treated with metformin, no treatment diabetic or have been treated but poorly balanced (HbA1c> 7%) and an applicant building with metformin; at any stage renal stable (stages 1-5 according to the classification MDRD)
* Patients aged 18 to 80 years;
* Patients with an assessment of renal function dating back more than 3 months;
* Patients whose renal function is stable, on the criterion of the absence of fluctuation over 30% of renal function of creatinine clearance in the last three months, a reference to renal function at least 3 months from the balance sheet inclusion is necessary.

Exclusion Criteria:

* Patient over 80 years
* Patients incapacitated adults (protected under guardianship)
* No previous reference creatinine;
* Fluctuation over 30% of renal function (creatinine clearance) in the three months;
* Reduction in BMI of more than 5% during the last 3 months;
* Severe hepatic impairment (Child stage> A);
* No reference to liver stages 3-5
* Patients to be an X-ray with injection of contrast.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
the percentage of patients in each category of renal function whose rate of erythrocyte metformin remain within the therapeutic range, at each stage of treatment. | Phase 1 : Day 7
the percentage of patients in each category of renal function whose rate of erythrocyte metformin remain within the therapeutic range, at each stage of treatment. | Phase 2 : Day 21
the percentage of patients in each category of renal function whose rate of erythrocyte metformin remain within the therapeutic range, at each stage of treatment. | Phase 3 : Day 35
the percentage of patients in stage 1 of chronic kidney disease (CKD) each category of renal function whose rate of erythrocyte metformin remain within the therapeutic range, at each stage of treatment. | Phase 4 : Day 49

SECONDARY OUTCOMES:
the percentage of patients in stages 3-5 of CKD each stage renal disease with a blood erythrocyte remaining within the therapeutic range or higher, and but without significative hyperlactatemia (≥ 2.5 mmol / l) in the latter case. | phase1 : Day 7
the percentage of patients in stages 3-5 of CKD each stage renal disease with a blood erythrocyte remaining within the therapeutic range or higher, and but without significative hyperlactatemia (≥ 2.5 mmol / l) in the latter case. | phase2 : Day 21
the percentage of patients in stages 3-5 of CKD each stage renal disease with a blood erythrocyte remaining within the therapeutic range or higher, and but without significative hyperlactatemia (≥ 2.5 mmol / l) in the latter case. | Phase3 : Day 35

CONTACTS AND LOCATIONS:
Overall Officials: LALAU J. Daniel, Professor, Principal Investigator — CHU Amiens
Locations (1):
- Service d'Endocrinologie, Maladies Métaboliques et Nutrition, Amiens, France

REFERENCES:
- [Result] Briet C, Saraval-Gross M, Kajbaf F, Fournier A, Hary L, Lalau JD. Erythrocyte metformin levels in patients with type 2 diabetes and varying severity of chronic kidney disease. Clin Kidney J. 2012 Feb;5(1):65-67. doi: 10.1093/ndtplus/sfr134. No abstract available. PMID 24596656